CLINICAL TRIAL: NCT04852250
Title: Impact of a Centralized Tumour Board on Secondary Intervention Rate in Patients With RAS Mutant Metastatic Colorectal Cancer After First-line Treatment With FOLFOXIRI Plus Bevacizumab (FIRE-7)
Brief Title: Centralized Tumour Board and Secondary Intervention Rate in mCRC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Charité Universitätsmedizin, Department of Hematology, Oncology and Tumor Immunology (Unknown)
Responsible Party: Principal Investigator, PD Dr. med. Volker Heinemann, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: FIRE-7
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Colorectal Cancer; RAS Mutation; Multidisciplinary Communication; Secondary Intervention
Keywords: metastatic colorectal cancer; RAS mutation; Multidisciplinary Communication; Secondary Intervention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FOLFOXIRI plus bevacizumab and centralized tumour board
  Interventions: Other: Virtual centralized multidisciplinary tumour board
- FOLFOXIRI plus bevacizumab but no centralized tumour board

INTERVENTIONS:
Other: Virtual centralized multidisciplinary tumour board — Evaluation of radiologic imaging and general condition by a multidisciplinary expert gremium to recommend either secondary intervention or resection of metastases or continuation of systemic treatment
  Groups: FOLFOXIRI plus bevacizumab and centralized tumour board

SUMMARY:
This is a randomised, multicentre observational study in patients suffering from RAS mutant mCRC with primarily unresectable metastases, who are planned to be treated with FOLFOXIRI and bevacizumab or who have already received ≤ four cycles FOLFOXIRI and bevacizumab as first-line treatment of metastatic disease. The patients are randomised in a 1:1 ratio to compare the rate of patients in whom secondary interventions (e.g. resection, ablation) are performed in curative intent when secondary intervention options are assessed by a multidisciplinary centralized tumour board (Arm A) versus when secondary intervention options are not assessed by a multidisciplinary centralized tumour board (Arm B).

All patients evaluated in the study will receive chemotherapy with FOLFOXIRI plus bevacizumab. After this induction/conversion therapy, imaging (CT or MRI) will be performed to evaluate resectability. In Arm A, a multidisciplinary, centralized tumour board will assess options of secondary intervention to be performed in the context of a generally curative treatment approach.

If there are secondary intervention options according to the judgement of the centralized tumour board, they will be listed in their respective sequence and the assessment will be communicated to the participating physician or his/her deputy at the study center. The decision, whether or not any secondary intervention is performed as recommended by the centralized tumour board as well as the kind of interventional procedures is up to the discretion of the treating physicians and surgeons of each patient. Any secondary intervention is recorded.

Evaluating the primary endpoint, the first interventions performed in one organ (e.g. liver) are rated when performed in a generally curative context (e.g. even in the presence of lung metastases that need to be approached in a further intervention).

In Arm B, no centralized tumour board will be integrated in to clinical decision making and patients will be treated according to institutional guidelines.

The number of treatment cycles with FOLFOXIRI and bevacizumab will be according to local clinical routine and medical guidelines, recommended are 8 to 12 cycles FOLFOXIRI in combination with bevacizumab, followed by a maintenance therapy with fluoropyrimidine (FP) plus bevacizumab until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study
2. Patients ≥ 18 years at the time of signing the informed consent
3. Histologically confirmed (in primary tumour or metastasis) UICC stage IV metastatic adenocarcinoma of the colon or rectum (mCRC) with primarily unresectable metastases
4. RAS mutant CRC (as determined by local pathology in tissue of primary tumour or metastasis)
5. At least one measurable lesion according to RECIST version 1.1 in a CT/MRI scan performed within 28 days prior to start of systemic treatment (first cycle of induction treatment)
6. ECOG performance status 0-1
7. Patients planned to receive chemotherapy with FOLFOXIRI plus bevacizumab as first-line treatment of metastatic disease. De-escalation of FOLFOXIRI to FOLFIRI or FOLFOX is allowed in case of toxicity.

   Patients can also be included if they had already received ≤ 4 cycles of induction/conversion therapy with FOLFOXIRI plus bevacizumab (including those patients in whom FOLFOXIRI has been de-escalated to FOLFIRI or FOLFOX due to toxicity) and the first restaging has not been conducted prior to randomization.
8. Completion of adjuvant therapy for colorectal cancer > 3 months prior to start of systemic treatment (first cycle of induction treatment).
9. Patient's ability for treatment with FOLFOXIRI and bevacizumab according to participating physician's judgement.

Exclusion Criteria:

1. Pregnant or breast-feeding women. Females of childbearing potential (FCBPs) who do not practice adequate contraceptive measures as required according to SmPCs of the administered medicinal products.
2. Contraindication to intensive chemotherapy with FOLFOXIRI plus bevacizumab
3. Contraindications to treatment with 5-FU, oxaliplatin, folinic acid, irinotecan (FOLFOXIRI) and/or bevacizumab according to SmPCs of the administered medicinal products.
4. Patients with confirmed cerebral metastasis. In case of clinical suspicion of brain metastasis, a cranial CT or MRI must be performed to rule out brain metastasis before study inclusion.
5. Documentation of > 5 lung metastases (however, no limitation for the number of metastases in the liver)
6. Isolated distant nodal metastasis, isolated peritoneal metastasis or isolated bone metastasis
7. Limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment naive patients with RAS mutated metastatic colorectal cancer who are planned to receive FOLFOXIRI plus bevacizumab or patients who already received up to 4 cycles of FOLFOXIRI plus bevacizumab.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Secondary intervention rate | 36 months
  Rate of patients in whom secondary interventions (e.g. resection, ablation treatment or combination of both) are performed in curative intent

SECONDARY OUTCOMES:
Objective response rate (ORR) according to RECIST 1.1 | 36 months
Progression-free survival (PFS) rate | 6, 12 and 16 months
Overall survival (OS) rate | 6, 12 and 16 months
Type, incidence, relatedness, and severity of adverse events with severity ≥ Grad 3 (severity according to NCI CTCAE version 5.0) | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, Prof., Principal Investigator — Ludwig-Maximilians - University of Munich

IPD SHARING:
Plan to Share IPD: No